CLINICAL TRIAL: NCT01517230
Title: Can Mass Media Campaigns Reduce Child Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Development Media International (Other); Centre Muraz (Other); Wellcome Trust (Other); Planet Wheeler Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-9-56; 6028 (Other: UK: Research ethics committee)
Record Dates: First submitted 2012-01-09; First posted 2012-01-25 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Diarrhoea; Malaria; Pneumonia; Breastfeeding; Under-nutrition
Keywords: Cluster-randomised trial; Comprehensive mass media campaign; Rural community radio; Under-five child mortality; Preventive and curative behaviours; Burkina Faso; Health care seeking behavior; Childbirth
MeSH Terms: conditions — Diarrhea; Malaria; Pneumonia; Breast Feeding; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Active Comparator): seven clusters where radio media campaign will be broadcast.
  Interventions: Behavioral: Local radio campaign to reduce under-five child mortality
- control (No Intervention): Seven clusters where radio media campaign won't be broadcast.

INTERVENTIONS:
Behavioral: Local radio campaign to reduce under-five child mortality — The media campaign is designed by Development Media International. It includes short "spots" and long format programs broadcast by rural community radios. Major topics to be addressed include: diarrhoea, water and sanitation, acute respiratory infections, fever/malaria, antenatal consultations, delivery in health facilities, breastfeeding, and child nutrition. The intervention is planned to start in March 2012 after completion of fieldwork for the baseline survey and will continue for 2.5 years.
  Arms: intervention

SUMMARY:
A cluster-randomised trial will be undertaken in Burkina Faso to investigate whether a comprehensive mass media campaign using local radio stations can change behaviours on a scale large enough to result in measurable and sustainable reductions in under-five child mortality.

It is hypothesised that as a result of the scale and multi-pronged nature of the campaign, reductions of between 10% and 20% in child mortality will be achieved.

DETAILED DESCRIPTION:
The evaluation is conducted in 14 geographical locations throughout Burkina Faso. Seven of these 14 clusters have been randomly allocated to receive the mass media intervention while the remaining 7 clusters will serve as controls.

Data collection includes household surveys in all 14 clusters at three "key" times:

* At baseline: Before the implementation of the intervention, between December 2011 and February 2012 to measure the current level of child mortality and evaluate current knowledge and behaviours of relevance to child health.
* At midline: Fifteen months after implementation of the intervention to evaluate the coverage of the intervention (in the intervention clusters) and, in each cluster, knowledge and behaviours.
* At endline: Two and a half years after implementation of the intervention to evaluate intervention coverage (in the intervention clusters), knowledge and behaviours and child mortality.

ELIGIBILITY:
Inclusion Criteria:

* Residence in study clusters

Exclusion Criteria:

* None

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100000 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Post neonatal under-five all cause mortality | 1 year

SECONDARY OUTCOMES:
Under-5 child all cause mortality | 1year
Preventive behaviours for main causes of under-five children mortality | 1 year
  1. Antenatal consultations during the last pregnancy which lasts more than 6 months and place of delivery
  2. Breastfeeding practices for the youngest under-five child
  3. Behaviours to prevent cases of diarrhoea and malaria in the youngest under-five child
Knowledge | 30-36 months after the start of the intervention
  1. Knowledge about danger signs during pregnancy, delivery and in young ill children
  2. Knowledge about preventive measure against malaria during pregnancy
  3. Knowledge about recommended breastfeeding behaviours
  4. Knowledge about transmission of malaria and diarrhoea
  5. Knowledge about health care seeking behaviours in young children suffering from diarrhoea, bad cough
Cost-effectiveness of mass media campaigns in terms of dollars per disability-adjusted life year (DALY) averted | 1 year
Curative behaviours for main causes of under-five children mortality | 15 days
  Health care behaviours to treat cases of diarrhoea, fever, cough and respiratory difficulties in the youngest under-five child during the 15 previous days

CONTACTS AND LOCATIONS:
Overall Officials: Simon N Cousens, MA, Principal Investigator — London School of Hygiene and Tropical Medicine; Nicolas Meda, MD, PhD, Principal Investigator — Centre Muraz; Sophie Sarrassat, PhD, Study Director — London School of Hygienne and Tropical Medicine; Moctar Ouedraogo, MsD, Study Director — Centre MURAZ / AfricSanté, Burkina Faso
Locations (1):
- Centre Muraz, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Kasteng F, Murray J, Cousens S, Sarrassat S, Steel J, Meda N, Ouedraogo M, Head R, Borghi J. Cost-effectiveness and economies of scale of a mass radio campaign to promote household life-saving practices in Burkina Faso. BMJ Glob Health. 2018 Jul 16;3(4):e000809. doi: 10.1136/bmjgh-2018-000809. eCollection 2018. PMID 30057798
- [Derived] Sarrassat S, Meda N, Badolo H, Ouedraogo M, Some H, Bambara R, Murray J, Remes P, Lavoie M, Cousens S, Head R. Effect of a mass radio campaign on family behaviours and child survival in Burkina Faso: a repeated cross-sectional, cluster-randomised trial. Lancet Glob Health. 2018 Mar;6(3):e330-e341. doi: 10.1016/S2214-109X(18)30004-4. PMID 29433668
- [Derived] Head R, Murray J, Sarrassat S, Snell W, Meda N, Ouedraogo M, Deboise L, Cousens S. Can mass media interventions reduce child mortality? Lancet. 2015 Jul 4;386(9988):97-100. doi: 10.1016/S0140-6736(14)61649-4. Epub 2015 Feb 13. PMID 25684587